CLINICAL TRIAL: NCT04115098
Title: Individualizing Anti-Inflammatory Medications for Adults With Axial Spondyloarthritis: A Series of N-of 1 Trials
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Mark C Hwang, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS-19-0677; KL2TR003168 (NIH)
Record Dates: First submitted 2019-10-02; First posted 2019-10-03 (Actual); Results first posted 2024-09-04 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Axial Spondyloarthritis
Keywords: spondylitis
MeSH Terms: conditions — Axial Spondyloarthritis; Spondylitis | interventions — Celecoxib; Naproxen; Meloxicam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (12):
- Celecoxib, Then Meloxicam, Then Naproxen, Then A, Then B (Experimental): Each participant will be randomized to a different initial drug sequence (6 possibilities: ABC, ACB, BAC, BCA, CBA, CAB) of the following three drugs: Naproxen 500 mg tablets twice daily (BID), Meloxicam 7.5 mg tablets BID and Celecoxib 200 mg capsules BID. After these 3 initial treatment sessions, participants are then randomized to the 2 best-performing drugs for 2 additional treatment sessions [randomized to either alphabetical order (A then B) or reverse alphabetical order (B then A)] There will be no washout periods. All 3 medications will be over-encapsulated in identical opaque capsules.
  Interventions: Drug: Celecoxib; Drug: Naproxen; Drug: Meloxicam
- Celecoxib, Then Meloxicam, Then Naproxen, Then B, Then A (Experimental): Each participant will be randomized to a different initial drug sequence (6 possibilities: ABC, ACB, BAC, BCA, CBA, CAB) of the following three drugs: Naproxen 500 mg tablets twice daily (BID), Meloxicam 7.5 mg tablets BID and Celecoxib 200 mg capsules BID. After these 3 initial treatment sessions, participants are then randomized to the 2 best-performing drugs for 2 additional treatment sessions [randomized to either alphabetical order (A then B) or reverse alphabetical order (B then A)] There will be no washout periods. All 3 medications will be over-encapsulated in identical opaque capsules.
  Interventions: Drug: Celecoxib; Drug: Naproxen; Drug: Meloxicam
- Celecoxib, Then Naproxen, Then Meloxicam, Then A, Then B (Experimental): Each participant will be randomized to a different initial drug sequence (6 possibilities: ABC, ACB, BAC, BCA, CBA, CAB) of the following three drugs: Naproxen 500 mg tablets twice daily (BID), Meloxicam 7.5 mg tablets BID and Celecoxib 200 mg capsules BID. After these 3 initial treatment sessions, participants are then randomized to the 2 best-performing drugs for 2 additional treatment sessions [randomized to either alphabetical order (A then B) or reverse alphabetical order (B then A)] There will be no washout periods. All 3 medications will be over-encapsulated in identical opaque capsules.
  Interventions: Drug: Celecoxib; Drug: Naproxen; Drug: Meloxicam
- Celecoxib, Then Naproxen, Then Meloxicam, Then B, Then A (Experimental): Each participant will be randomized to a different initial drug sequence (6 possibilities: ABC, ACB, BAC, BCA, CBA, CAB) of the following three drugs: Naproxen 500 mg tablets twice daily (BID), Meloxicam 7.5 mg tablets BID and Celecoxib 200 mg capsules BID. After these 3 initial treatment sessions, participants are then randomized to the 2 best-performing drugs for 2 additional treatment sessions [randomized to either alphabetical order (A then B) or reverse alphabetical order (B then A)] There will be no washout periods. All 3 medications will be over-encapsulated in identical opaque capsules.
  Interventions: Drug: Celecoxib; Drug: Naproxen; Drug: Meloxicam
- Meloxicam, Then Celecoxib, Then Naproxen, Then A, Then B (Experimental): Each participant will be randomized to a different initial drug sequence (6 possibilities: ABC, ACB, BAC, BCA, CBA, CAB) of the following three drugs: Naproxen 500 mg tablets twice daily (BID), Meloxicam 7.5 mg tablets BID and Celecoxib 200 mg capsules BID. After these 3 initial treatment sessions, participants are then randomized to the 2 best-performing drugs for 2 additional treatment sessions [randomized to either alphabetical order (A then B) or reverse alphabetical order (B then A)] There will be no washout periods. All 3 medications will be over-encapsulated in identical opaque capsules.
  Interventions: Drug: Celecoxib; Drug: Naproxen; Drug: Meloxicam
- Meloxicam, Then Celecoxib, Then Naproxen, Then B, Then A (Experimental): Each participant will be randomized to a different initial drug sequence (6 possibilities: ABC, ACB, BAC, BCA, CBA, CAB) of the following three drugs: Naproxen 500 mg tablets twice daily (BID), Meloxicam 7.5 mg tablets BID and Celecoxib 200 mg capsules BID. After these 3 initial treatment sessions, participants are then randomized to the 2 best-performing drugs for 2 additional treatment sessions [randomized to either alphabetical order (A then B) or reverse alphabetical order (B then A)] There will be no washout periods. All 3 medications will be over-encapsulated in identical opaque capsules.
  Interventions: Drug: Celecoxib; Drug: Naproxen; Drug: Meloxicam
- Meloxicam, Then Naproxen, Then Celecoxib, Then A, Then B (Experimental): Each participant will be randomized to a different initial drug sequence (6 possibilities: ABC, ACB, BAC, BCA, CBA, CAB) of the following three drugs: Naproxen 500 mg tablets twice daily (BID), Meloxicam 7.5 mg tablets BID and Celecoxib 200 mg capsules BID. After these 3 initial treatment sessions, participants are then randomized to the 2 best-performing drugs for 2 additional treatment sessions [randomized to either alphabetical order (A then B) or reverse alphabetical order (B then A)] There will be no washout periods. All 3 medications will be over-encapsulated in identical opaque capsules.
  Interventions: Drug: Celecoxib; Drug: Naproxen; Drug: Meloxicam
- Meloxicam, Then Naproxen, Then Celecoxib, Then B, Then A (Experimental): Each participant will be randomized to a different initial drug sequence (6 possibilities: ABC, Each participant will be randomized to a different initial drug sequence (6 possibilities: ABC, ACB, BAC, BCA, CBA, CAB) of the following three drugs: Naproxen 500 mg tablets twice daily (BID), Meloxicam 7.5 mg tablets BID and Celecoxib 200 mg capsules BID. After these 3 initial treatment sessions, participants are then randomized to the 2 best-performing drugs for 2 additional treatment sessions [randomized to either alphabetical order (A then B) or reverse alphabetical order (B then A)] There will be no washout periods. All 3 medications will be over-encapsulated in identical opaque capsules.
  Interventions: Drug: Celecoxib; Drug: Naproxen; Drug: Meloxicam
- Naproxen, Then Celecoxib, Then Meloxicam, Then A, Then B (Experimental): Each participant will be randomized to a different initial drug sequence (6 possibilities: ABC, ACB, BAC, BCA, CBA, CAB) of the following three drugs: Naproxen 500 mg tablets twice daily (BID), Meloxicam 7.5 mg tablets BID and Celecoxib 200 mg capsules BID. After these 3 initial treatment sessions, participants are then randomized to the 2 best-performing drugs for 2 additional treatment sessions [randomized to either alphabetical order (A then B) or reverse alphabetical order (B then A)] There will be no washout periods. All 3 medications will be over-encapsulated in identical opaque capsules.
  Interventions: Drug: Celecoxib; Drug: Naproxen; Drug: Meloxicam
- Naproxen, Then Celecoxib, Then Meloxicam, Then B, Then A (Experimental): Each participant will be randomized to a different initial drug sequence (6 possibilities: ABC, ACB, BAC, BCA, CBA, CAB) of the following three drugs: Naproxen 500 mg tablets twice daily (BID), Meloxicam 7.5 mg tablets BID and Celecoxib 200 mg capsules BID. After these 3 initial treatment sessions, participants are then randomized to the 2 best-performing drugs for 2 additional treatment sessions [randomized to either alphabetical order (A then B) or reverse alphabetical order (B then A)] There will be no washout periods. All 3 medications will be over-encapsulated in identical opaque capsules.
  Interventions: Drug: Celecoxib; Drug: Naproxen; Drug: Meloxicam
- Naproxen, Then Meloxicam, Then Celecoxib, Then A, Then B (Experimental): Each participant will be randomized to a different initial drug sequence (6 possibilities: ABC, ACB, BAC, BCA, CBA, CAB) of the following three drugs: Naproxen 500 mg tablets twice daily (BID), Meloxicam 7.5 mg tablets BID and Celecoxib 200 mg capsules BID. After these 3 initial treatment sessions, participants are then randomized to the 2 best-performing drugs for 2 additional treatment sessions [randomized to either alphabetical order (A then B) or reverse alphabetical order (B then A)] There will be no washout periods. All 3 medications will be over-encapsulated in identical opaque capsules.
  Interventions: Drug: Celecoxib; Drug: Naproxen; Drug: Meloxicam
- Naproxen, Then Meloxicam, Then Celecoxib, Then B, Then A (Experimental): Each participant will be randomized to a different initial drug sequence (6 possibilities: ABC, ACB, BAC, BCA, CBA, CAB) of the following three drugs: Naproxen 500 mg tablets twice daily (BID), Meloxicam 7.5 mg tablets BID and Celecoxib 200 mg capsules BID. After these 3 initial treatment sessions, participants are then randomized to the 2 best-performing drugs for 2 additional treatment sessions [randomized to either alphabetical order (A then B) or reverse alphabetical order (B then A)] There will be no washout periods. All 3 medications will be over-encapsulated in identical opaque capsules.
  Interventions: Drug: Celecoxib; Drug: Naproxen; Drug: Meloxicam

INTERVENTIONS:
Drug: Celecoxib — Celecoxib 200 mg capsules twice daily (BID) All 3 medications will be over-encapsulated in identical opaque capsules
Drug: Naproxen — Naproxen 500 mg tablets twice daily (BID) All 3 medications will be over-encapsulated in identical opaque capsules
Drug: Meloxicam — Meloxicam 7.5 mg tablets twice daily (BID) All 3 medications will be over-encapsulated in identical opaque capsules

SUMMARY:
The purpose of this study is to compare selective cyclooxygenase-2 (COX-2) and non selective COX inhibitors with respect to the extent to which disease activity is improved without self reported, unacceptable side effects among individual patients with axial spondyloarthritis (AxSpA),to compare selective COX-2 and nonselective COX inhibitors impact on Health related Quality of Life (HrQOL) and how this relates to changes in disease activity and to conduct proteomic assessment of predictive biomarkers of non steroidal anti-inflammatory drug(NSAID) response

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet modified New York Classification and/or Assessment of Spondyloarthritis International Society (ASAS) criteria for Classification Criteria for AxSpA
* Ankylosing Spondylitis Disease Activity Score greater than or equal to 2.1.

Exclusion Criteria:

* Changing background biologic/disease modifying-rheumatic medications within less than 3 months.
* Opioid medication use
* Current or expected pregnancy
* History of cardiovascular disease (previous stroke, myocardial infarction, or percutaneous intervention.
* End stage liver disease
* Chronic Kidney Disease greater than Stage IIIb

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark C Hwang, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hwang MC, Kim S, Assassi S, Chavez R, Samuel J, Green C, Tyson J, Reveille J. Individualizing NSAID therapy in axial spondyloarthritis: N-of-1 trials with Bayesian analysis. Rheumatology (Oxford). 2025 Dec 1;64(12):6114-6121. doi: 10.1093/rheumatology/keaf393. PMID 40676732

RESULTS

PARTICIPANT FLOW:
Groups:
- Meloxicam, Then Naproxen, Then Celecoxib, Then B, Then A; Naproxen, Then Celecoxib, Then Meloxicam, Then A, Then B; Naproxen, Then Celecoxib, Then Meloxicam, Then B, Then A; Naproxen, Then Meloxicam, Then Celecoxib, Then A, Then B; Naproxen, Then Meloxicam, Then Celecoxib, Then B, Then A: Each participant will be randomized to a different initial drug sequence (6 possibilities: ABC, ACB, BAC, BCA, CBA, CAB) of the following three drugs: Naproxen 500 mg tablets twice daily (BID), Meloxicam 7.5 mg tablets BID and Celecoxib 200 mg capsules BID. After these 3 initial treatment sessions, participants are then randomized to the 2 best-performing drugs for 2 additional treatment sessions [randomized to either alphabetical order (A then B) or reverse alphabetical order (B then A)] There will be no washout periods. All 3 medications will be over-encapsulated in identical opaque capsules.
Period: Overall Study
Arm/Group | Celecoxib, Then Meloxicam, Then Naproxen, Then A, Then B | Celecoxib, Then Meloxicam, Then Naproxen, Then B, Then A | Celecoxib, Then Naproxen, Then Meloxicam, Then A, Then B | Celecoxib, Then Naproxen, Then Meloxicam, Then B, Then A | Meloxicam, Then Celecoxib, Then Naproxen, Then A, Then B | Meloxicam, Then Celecoxib, Then Naproxen, Then B, Then A | Meloxicam, Then Naproxen, Then Celecoxib, Then A, Then B | Meloxicam, Then Naproxen, Then Celecoxib, Then B, Then A | Naproxen, Then Celecoxib, Then Meloxicam, Then A, Then B | Naproxen, Then Celecoxib, Then Meloxicam, Then B, Then A | Naproxen, Then Meloxicam, Then Celecoxib, Then A, Then B | Naproxen, Then Meloxicam, Then Celecoxib, Then B, Then A
Started | 5 | 2 | 3 | 4 | 5 | 2 | 0 | 7 | 4 | 3 | 4 | 3
4-week Treatment Session 1 | 5 | 2 | 3 | 4 | 5 | 2 | 0 | 7 | 4 | 3 | 4 | 3
4-week Treatment Session 2 | 4 | 2 | 3 | 4 | 4 | 2 | 0 | 6 | 3 | 3 | 4 | 3
4-week Treatment Session 3 | 3 | 2 | 3 | 4 | 4 | 1 | 0 | 6 | 3 | 2 | 4 | 2
4-week Treatment Session 4 | 3 | 2 | 3 | 4 | 3 | 1 | 0 | 6 | 2 | 2 | 4 | 2
4-week Treatment Session 5 | 2 | 2 | 3 | 4 | 3 | 1 | 0 | 6 | 2 | 1 | 4 | 2
Completed | 2 | 2 | 3 | 4 | 3 | 1 | 0 | 6 | 2 | 1 | 4 | 2
Not Completed | 3 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 2 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Each participant will be randomized to a different initial drug sequence (6 possibilities: ABC, ACB, BAC, BCA, CBA, CAB) of the following three drugs: Naproxen 500 mg tablets twice daily (BID), Meloxicam 7.5 mg tablets BID and Celecoxib 200 mg capsules BID. After these 3 initial treatment sessions, participants are then randomized to the 2 best-performing drugs for 2 additional treatment sessions [randomized to either alphabetical order (A then B) or reverse alphabetical order (B then A)] There will be no washout periods. All 3 medications will be over-encapsulated in identical opaque capsules.
Arm/Group | All Participants
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.40 (13)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex data were not collected from any participant.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Disease Activity as Measured by the Ankylosing Spondylitis Disease Activity Score (ASDAS)
Description: The ASDAS total score ranges from 0-10, with a higher score meaning worse disease activity. The change in score is reported as [(ASDAS score at baseline) - (ASDAS score at 4 weeks)]--a positive value indicates that the score (and disease activity) decreased over time.
  The "Measure of Dispersion/Precision" indicated as "95% Confidence Interval" actually refers to a "95% Credible Interval."
Time Frame: Baseline, 4 weeks
Measure: Median (95% Confidence Interval); unit: score on a scale
Groups:
- Celecoxib: Celecoxib 200 mg capsules BID
- Meloxicam: Meloxicam 7.5 mg tablets
- Naproxen: Naproxen 500 mg tablets twice daily (BID)
Arm/Group | Celecoxib | Meloxicam | Naproxen
Number analyzed (Participants) | 30 | 30 | 30
score on a scale | 0.61 [0.35 to 0.87] | 0.54 [0.28 to 0.81] | 0.58 [0.32 to 0.84]

2. Secondary Outcome: Change in Health Related Quality of Life as Assessed by the Standard Gamble Utility Assessment
Description: The Standard Gamble Utility assessment is scored between 0-1, with 0 being the worst outcome and 1 being the best outcome. The change in score is reported as [(Standard Gamble score at baseline) - (Standard Gamble score at 4 weeks)]--a negative value indicates that the Health Related Quality of Life increased over time. The "Measure of Dispersion/Precision" indicated as "95% Confidence Interval" actually refers to a "95% Credible Interval.
Time Frame: Baseline, 4 weeks
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Celecoxib | Meloxicam | Naproxen
Number analyzed (Participants) | 30 | 30 | 30
score on a scale | -0.07 [-0.18 to 0.04] | -0.04 [-0.16 to 0.07] | -0.05 [-0.16 to 0.06]

3. Secondary Outcome: Change in Health-Related Quality of Life as Assessed by the PROMIS-Preference (PROPr) Score
Description: The reported Patient-Reported Outcomes Measurement Information System-Preference (PROPr) Score ranges from 0 to 1, with 0 being the worst outcome and 1 being the best outcome. The change in score is reported as [(PROPr score at baseline) - (PROPR score at 4 weeks)] - a negative value indicates that the person's Health Related Quality of Life increased over time. The "Measure of Dispersion/Precision" indicated as "95% Confidence Interval" actually refers to a "95% Credible Interval."
Time Frame: Baseline, 4 weeks
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Celecoxib | Meloxicam | Naproxen
Number analyzed (Participants) | 30 | 30 | 30
score on a scale | -0.10 [-0.14 to -0.05] | -0.11 [-0.16 to -0.06] | -0.11 [-0.16 to -.06]

4. Secondary Outcome: Change in Ability to Perform Tasks as Assessed by the Bath Ankylosing Spondylitis Functional Index (BASFI)
Description: BASFI score ranges from 0-10, with 0 being easy and 10 being impossible. The change in score is reported as [(BASFI score at baseline) - (BASFI score at 4 weeks)], and a positive value indicates that the score (and difficulty with tasks) decreased over time.
  The "Measure of Dispersion/Precision" indicated as "95% Confidence Interval" actually refers to a "95% Credible Interval."
Time Frame: Baseline, 4 weeks
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Celecoxib | Meloxicam | Naproxen
Number analyzed (Participants) | 30 | 30 | 30
score on a scale | 0.55 [0.11 to 1] | 0.53 [0.08 to 0.99] | 0.37 [-0.07 to 0.83]

5. Secondary Outcome: Change in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)
Description: The BASDAI consists of a 0 - 10 scale measuring discomfort, pain, and fatigue (0 being no problem and 10 being the worst problem). The change in score is reported as [(BASDAI score at baseline) - (BASDAI score at 4 weeks)] -- a positive value indicates that the score (and disease activity) decreased over time. The "Measure of Dispersion/Precision" indicated as "95% Confidence Interval" actually refers to a "95% Credible Interval."
Time Frame: Baseline, 4 weeks
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Celecoxib | Meloxicam | Naproxen
Number analyzed (Participants) | 30 | 30 | 30
score on a scale | 1.07 [0.49 to 1.63] | 1.19 [0.62 to 1.76] | 1.17 [0.59 to 1.74]

6. Secondary Outcome: Change in Bath Ankylosing Spondylitis Metrology Index (BASMI)
Description: BASMI total score ranges from 0 - 10.The higher the BASMI score, the more severe the patient's limitation of movement due to their ankylosing spondylitis. The change in score is reported as [(BASMI score at baseline) - (BASMI score at 4 weeks)]--a positive value indicates that the score (and limitation of movement) decreased over time.
  The "Measure of Dispersion/Precision" indicated as "95% Confidence Interval" actually refers to a "95% Credible Interval."
Time Frame: Baseline, 4 weeks
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Celecoxib | Meloxicam | Naproxen
Number analyzed (Participants) | 30 | 30 | 30
score on a scale | 0.15 [-0.07 to 0.37] | 0.03 [-0.19 to 0.26] | 0.11 [-0.11 to 0.33]

7. Secondary Outcome: Change in Pain as Assessed by the Visual Analog Scale-Pain (VAS-Pain)
Description: The VAS-Pain total score is 0 - 100, with 0 being no pain and 100 being unbearable pain. The change in score is reported as [(VAS- Pain score at baseline) - (VAS- Pain score at 4 weeks)] --a positive value indicates that the score (and pain level) decreased over time. The "Measure of Dispersion/Precision" indicated as "95% Confidence Interval" actually refers to a "95% Credible Interval."
Time Frame: Baseline, 4 weeks
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Celecoxib | Meloxicam | Naproxen
Number analyzed (Participants) | 30 | 30 | 30
score on a scale | 11.28 [5.32 to 17.22] | 11.26 [5.26 to 17.18] | 11.32 [5.42 to 17.12]

8. Secondary Outcome: Change in Visual Analog Scale-Global (VAS-Global)
Description: The VAS-Global is scored from 0-100, with 0 being not active and 100 being very active. The change in score is reported as [(VAS- Global score at baseline) - (VAS- Global score at 4 weeks)] --a negative value indicates that the score (and activity level) increased over time. The "Measure of Dispersion/Precision" indicated as "95% Confidence Interval" actually refers to a "95% Credible Interval."
Time Frame: Baseline, 4 weeks
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Celecoxib | Meloxicam | Naproxen
Number analyzed (Participants) | 30 | 30 | 30
score on a scale | 14.29 [7.94 to 20.35] | 14.33 [7.97 to 20.38] | 14.39 [8.13 to 20.36]

ADVERSE EVENTS:
Time Frame: 29 weeks
Groups:
- Celecoxib: Celecoxib 200 mg capsules twice daily (BID)
- Meloxicam: Meloxicam 7.5 mg tablets twice daily (BID)
Arm/Group | Celecoxib | Meloxicam | Naproxen
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 1/30 | 0/30
Other Adverse Events (participants affected / at risk) | 2/30 | 4/30 | 5/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Celecoxib (N=30) | Meloxicam (N=30) | Naproxen (N=30)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Celecoxib (N=30) | Meloxicam (N=30) | Naproxen (N=30)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomach Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (11)

LIMITATIONS AND CAVEATS:
Terminated due to lack of recruitment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-16): https://cdn.clinicaltrials.gov/large-docs/98/NCT04115098/Prot_SAP_000.pdf